CLINICAL TRIAL: NCT03223090
Title: A Motor Tool for Language Learning
Brief Title: Motor Language Learning
Acronym: MOTOLANGUAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 69HCL17_0359; 2017-A02144-49 (Other: ID-RCB)
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Language; learning; plasticity
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tool training group (Experimental): Motor training with a tool during max 5 weeks (3 days per week, around 30 minutes per day)
  Interventions: Behavioral: Tool-use
- Hand training group (Active Comparator): Motor training with the right hand during max 5 weeks (3 days per week, around 30 minutes per day)
  Interventions: Behavioral: Hand

INTERVENTIONS:
Behavioral: Tool-use — Motor training with a tool during max 5 weeks (3 days per week, around 30 minutes per day)
  Arms: Tool training group
Behavioral: Hand — Motor training with the right hand during max 5 weeks (3 days per week, around 30 minutes per day)
  Arms: Hand training group

SUMMARY:
This project pursues the validation of an innovative strategy to boost language learning, based on the benefits derived from sensorimotor training.

The common belief of a rigid brain structure in adult life had to be reconsidered during the last decade. After training, local increase in cerebral cortex volume and thickness, the part of the brain containing neuronal cells and synapses, has been documented. Research has established that brain structures active during training expand while learning and return to baseline afterwards. The transient structural increase is thought to reflect "work in progress" within areas involved in learning, meant to integrate new skills in existing neural circuitries, via strengthening and/or selection of local neuronal connections. My main hypothesis is that other functions, as long as they rely on the activity of the same brain territories, can take advantage of this "work in progress". To use an allegory, imagine the restauration of a building (brain area). It can start after the request of improvements from some of the residents (trained function) and then become the occasion for other tenants (other functions) to see realized also their own wish for improvements. In the end everybody will benefit from the restauration, provided that they all live in the same building and everybody has posed their requests during the "work in progress". Out of the allegory, living in the same building means neural overlap of functions in the brain. The case of motor and linguistic systems represents, from this perspective, a unique opportunity. State-of-the-art research 1) proved the existence, and described the temporal evolution of brain plastic changes during sensorimotor learning, and 2) documented neural overlap and functional interactions of motor and linguistic systems. This posits solid bases for a crucial step forward, gravid of important consequences and applications. This project aims to take this step forward by directly testing the innovative hypothesis that brain changes induced by sensorimotor learning induce benefits for linguistic functions relying on the same brain territories.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 20 and 40 years old
* Give an informed consent by signature
* Be part of the national health security system (registered to the Securité Sociale)
* Be French speaker

Exclusion Criteria:

* A person presenting an history of neurological, psychiatric or linguistic problems cannot be admitted
* Assumption of psychotropic drugs
* Pregnancy or breast-feeding woman
* A person under legal tutoring
* A person under care in other medical structure for reasons different from those of this research
* A person under administrative or judiciary contention
* A person who is not eligible to a MR-exam according to the relative screening questionnaire cannot be admitted to the experiments including MR acquisitions in the protocol
* A person who is not eligible to a tDC Stimulation according to the relative screening questionnaire cannot be admitted to the experiment including tDCS in the protocol
* A person who is defined as bilingual according to the criteria described above cannot be included in this research.
* A person who studied a musical instrument for more than 3 years or plays it regularly cannot take part to the studies in Objective B1, B2 and B3. This might introduce a confound in the rate of motor learning and relative brain plasticity.
* A person who has already learned or has been regularly exposed to the language L2 and/or to the sign language chosen for the studies in Objective A1 and A2 cannot take part to those studies.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1111 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2027-03-19 (Estimated); Study Completion 2027-03-19 (Estimated)

PRIMARY OUTCOMES:
Linguistic performance amelioration ratio | max 6 weeks after motor training started
  (Post Accuracy % - Pre Accuracy %) and/or (Pre RTs (ms) - Post RTs (ms))

CONTACTS AND LOCATIONS:
Overall Officials: Claudio BROZZOLI, Principal Investigator — INSERM U1028 - Impact - CRNL
Locations (1):
- Hospices Civils de Lyon, Bron, France